CLINICAL TRIAL: NCT03507634
Title: Opioid Free Anesthesia in Bariatric Surgery: A Prospective, Double-blinded, Randomized, Controlled Clinical Trial
Brief Title: Opioid Free Anesthesia in Bariatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lebanese American University (Other)
Responsible Party: Principal Investigator, Hanane Barakat, MD, Lebanese American University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LAUMCRH.HB2.28/Mar/2018
Record Dates: First submitted 2018-04-12; First posted 2018-04-25 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Opioid Use; Postoperative Pain; Postoperative Nausea and Vomiting; Bariatric Surgery Candidate
Keywords: Lidocaine; Dexmedetomidine; Opioid Free; Bariatric surgery
MeSH Terms: conditions — Pain, Postoperative; Postoperative Nausea and Vomiting | interventions — Lidocaine; Remifentanil

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Opioid Based Anesthesia (Active Comparator): General anesthesia will be induced using Propofol , fentanyl , and Rocuronium . Ketamine will be administered on induction of anesthesia with the same dose to be repeated every hour. Anesthesia will be maintained with Remi-fentanyl and Sevoflurane.
  Interventions: Drug: Opioid based anesthesia Fentanyl and Remifentanyl
- Opioid Free Anesthesia (Active Comparator): General anesthesia will be induced using dexmedetomidine and lidocaine started 10 minutes before induction, Propofol and Rocuronium . Ketamine will be administered on induction of anesthesia with the same dose to be repeated every hour. Anesthesia will be maintained with IV infusion of dexmedetomidine , lidocaine and Sevoflurane.
  Interventions: Drug: Opioid free Anesthesia dexmedetomidine and lidocaine

INTERVENTIONS:
Drug: Opioid free Anesthesia dexmedetomidine and lidocaine — Opioid free anesthesia with dexmedetomidine and lidocaine
  Arms: Opioid Free Anesthesia
Drug: Opioid based anesthesia Fentanyl and Remifentanyl — Opioid based anesthesia with Fentanyl and Remifentanyl
  Arms: Opioid Based Anesthesia

SUMMARY:
This study compares the intraoperative opioid free anesthesia approach in laparoscopic bariatric surgery to a conventional opioid- based anesthesia. Half of participants will receive opioid free anesthesia with dexmedetomidine, lidocaine and ketamine while the other half will receive opioid based anesthesia with fentanyl, remi-fentanyl and ketamine

DETAILED DESCRIPTION:
Since optimal analgesia for the obese patients undergoing bariatric surgeries has always been challenging, and knowing the comorbidities and physiological changes in this population, use of opioid-sparing agents during anesthesia has attracted substantial research.the use of opioids in the perioperative period in obese patients is associated with an increased risk of complications . They are especially more sensitive to the respiratory depressant effect of opioids , thus any analgesic alternative without further compromising airway tone would be a desirable choice.

Dexmedetomidine is a selective alpha-two adrenergic receptor agonist that has antinociceptive, analgesic and sedative properties, without compromising airway tone and reflexes .

Lidocaine, a local anesthetic that has been shown to be an effective multimodal strategy to minimize postoperative pain was evaluated in one study involving obese patients undergoing bariatric surgery. Its usage was associated with an improved quality of recovery compared to placebo .

ELIGIBILITY:
Inclusion Criteria:

* Age group: 18-65 years old
* American Society of Anesthesiologists (ASA )class I and II
* Indicated laparoscopic bariatric surgery

Exclusion Criteria:

* Renal, hepatic or cardiac insufficiency
* Positive pregnancy test
* Alcohol or drug abuse
* Psychiatric disease
* History of chronic pain
* Allergy or contraindication to any of the study drugs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-04-11 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Postoperative pain score for 48 hours | 48 hours postoperative
  Measure the pain score using the Visual Analogue Scale (VAS), The Visual Analogue Scale (VAS) consists of a straight line with the endpoints defining extreme limits such as 'no pain at all' and 'pain as bad as it could be' The patient is asked to mark his pain level on the line between the two endpoints. The distance between 'no pain at all' and the mark then defines the subject's pain. The score ranges from 0 to 100 mm. A higher score indicates greater pain intensity. The distribution pain is the following:no pain (0-4 mm), mild pain(5-44 mm), moderate pain (45-74 mm), and severe pain (75-100 mm).Postoperative pain will be measured using Verbal Analogue Scale (VAS) at 0, 1, 2, 4, 6, 12, 18, and 24 and every 6 hours up to 48 hours post surgery.

SECONDARY OUTCOMES:
Postoperative morphine consumption at the PACU (Post Anesthesia Care Unit) | 2 hours postoperative
  After the surgery the patient will go to the PACU (Post Anesthesia Care Unit). the patient will receive morphine if the pain score is more than 4. the total dose of morphine in mg (milligrams) will be documented.
Postoperative morphine consumption at the surgical ward for 48 hours | 48 hours postoperative
  Post-operative opioid consumption will be based on the amount in mg (milligrams) of opioid required in the 48 hours postoperative.
Postoperative morphine Side effects: Sedation score .for 48 hours | 48 hours postoperative
  Sedation score:
  0 alert
  1. Mild, drowsy , easy to awake
  2. moderate, easy to arouse
  3. Severe: somnolent difficult to arouse 4:sleeping The Sedation score will be documented at 0, 1, 2, 4, 6, 12, 18, and 24 hours and then every 6 hours up to 48 hours.
Postoperative morphine Side effects:Respiratory depression for 48 hours | 48 hours postoperative
  Assess the respiratory rate : The number of breaths per minute. In practice, the respiratory rate is usually determined by counting the number of times the chest rises or falls per minute.
  The respiratory rate will be documented at 0, 1, 2, 4, 6, 12, 18, and 24 hours and then every 6 hours up to 48 hours.
Postoperative morphine Side effects: Nausea vomiting for 48 hours | 48 hours postoperative
  Degree of nausea vomiting using the verbal rating score from 0 to 10 :
  0= no nausea/ Vomiting, 10: worst possible nausea vomiting.
  The degree of nausea vomiting will be documented at 0, 1, 2, 4, 6, 12, 18, and 24 hours and every 6 hours thereafter up to 48 hours.
Postoperative morphine Side effects: Itching for 48 hours | 48 hours postoperative
  Itching: presence or absence The presence or absence of itching will be documented at 0, 1, 2, 4, 6, 12, 18, and 24 hours and every 6 hours thereafter up to 48 hours.

CONTACTS AND LOCATIONS:
Locations (1):
- LAU Medical Center, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Barakat H, Gholmieh L, Nader JA, Karam VY, Albaini O, Helou ME, Al Nawwar R. Opioid-free versus opioid-based anesthesia in laparoscopic sleeve gastrectomy: a single-center, randomized, controlled trial. Perioper Med (Lond). 2025 Feb 5;14(1):16. doi: 10.1186/s13741-024-00486-5. PMID 39910664